CLINICAL TRIAL: NCT04244149
Title: Exploring the Effect of Exhaustive Exercise From a Metabolomic and Metagenomic Approach
Brief Title: Effect of an Exercise Bout in Plasma and Fecal Profile
Acronym: MEMEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Mar Larrosa, Tenure Professor, Universidad Europea de Madrid
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UEM0003
Record Dates: First submitted 2020-01-20; First posted 2020-01-28 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Participants will exert an exercise prolonged session
  Interventions: Other: Prolonged Exercise session

INTERVENTIONS:
Other: Prolonged Exercise session — After a standardized warm-up of 10 minutes of continuous running on a treadmill at 60% of their maximum heart rate (HRmax), subjects will perform a maximum oxygen consumption test (VO2max) with a gas analyzer (UltimaTM Series, MGC Diagnostic Corporation, St. Paul, MN, USA. The protocol will start with a slope of 1% at a speed of 10 km/h, with increments of 0.3 km/h every 30 s until volitional exhaustion. Finally, ten minutes after the treadmill test, volunteers will run 1 kilometer (t1km) as fast as possible and the time needed to cover the distance will be recorded.

SUMMARY:
The aim of this project is to study the effect of a bout of exercise on the metabolomic profile of plasma and feces as well as its influence on the intestinal microbiota.

DETAILED DESCRIPTION:
The practice of physical exercise has numerous health benefits, preventing the appearance and development of cardiovascular diseases and various types of cancer. Exercise causes changes in the vascular, muscular and pulmonary systems, etc. One of the benefits that can result from exercise modification of the intestinal microbiota and its metabolic profile. In order to identify the potential changes that exercise has on the intestinal microbiota and its metabolic profile, the purpose of this study is to identify changes in the plasma and fecal metabolome and in fecal microbiota associated with a bout of exercise

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years of age
* high physical condition (VO2 ≥ 55 ml/kg/min)
* BMI 18-25 kg/m2

Exclusion Criteria:

* antibiotics intake during 3 months prior to the study,
* smoking
* nutritional complements
* ergogenic complements
* prebiotics
* probiotics
* vegetarian or vegan diet
* chronic medication
* gastrointestinal surgery
* Any diagnosed disease

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Plasma metabolome profile | Changes from baseline to 30 min after the exercise intervention
  Abundance of blood metabolites, metabolic networks, and metabolic pathways activity
Fecal microbiota | Changes from baseline to 30 min after the exercise intervention
  Abundance of gut microbial taxa, communities, and metabolic pathways activity

CONTACTS AND LOCATIONS:
Overall Officials: Mar Larrosa, PhD, Principal Investigator — Universidad Europea de Madrid
Locations (1):
- Maria del Mar Larrosa Pérez, Villaviciosa de Odón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication. Metagenomic raw data will be deposited in the http://www.ncbi.nlm.nih.gov/sra
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Upon publication
Access Criteria: Data will be in a public repository